CLINICAL TRIAL: NCT02983279
Title: Caloric Restriction for Oncology Research: Pre-operative Caloric Restriction Prior to Definitive Oncologic Surgery
Brief Title: Caloric Restriction Before Surgery in Treating Patients With Endometrial, Prostate, or Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16D.501; JT 8646 (Other: JeffTrial Number)
Record Dates: First submitted 2016-11-14; First posted 2016-12-06 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Carcinoma; Endometrial Carcinoma; Prostate Carcinosarcoma
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms | interventions — Diet Therapy; Counseling; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dietary counseling, caloric restriction diet (Experimental): Patients then undergo 25% caloric intake for 3-12 weeks prior to definitive cancer surgery.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Counseling; Procedure: Therapeutic

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Undergo caloric restriction diet
  Other Names: Dietary Modification; Nutrition Intervention
Other: Counseling — Undergo counselor-led dietary counseling
  Other Names: Counseling Intervention
Procedure: Therapeutic — Undergo standard of care surgery

SUMMARY:
The purpose of this trial is to determine that sort term calorie restriction will affect tumor biology in biopsy proven breast, endometrial or prostate cancers, which will positively impact biomarkers including miR-21, an onco-miR known to impact cancer outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1) Investigate if caloric restriction will change serum micro ribonucleic acid (RNA) 21 (miR-21) expression in patients with prostate, endometrial or breast cancer.

SECONDARY OBJECTIVES:

1. Investigate measurable changes induced by caloric restriction on both patient (host) and tumor characteristics from caloric restriction.
2. Investigate the adherence of the patient to the diet.

4) Weight, height, and body composition will be assessed via BodyMetrix. BodyMetrix uses ultrasound technology to measure subcutaneous fat.

5) Patients will have psycho-social evaluation using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) test (prostate cancer), FACT-Breast (B) test (breast cancer), or the FACT-Endometrial Cancer (En) test (endometrial cancer) and the Patient Reported Outcomes Measurement Information System (PROMIS) cancer fatigue short form at baseline, midway through diet, and at the conclusion of the diet.

6) Patient's nutritional status (Mini Nutritional Assessment [MNA] form) will be assessed, and their caloric needs will be calculated.

7) Local recurrence, progression free survival, distant metastases and overall survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Histological documentation of cancer of the endometrium, prostate or breast.
2. Candidate for definitive cancer surgery as determined by treating physician
3. The ability for the definitive cancer surgery to be scheduled within 4-12 weeks post initiation of dietary intervention as determined by the enrolling physician (not from diagnosis - but from start of diet).
4. No other malignancy within the past 6 months unless it was a non-melanomatous skin lesion
5. BMI ≥21
6. ECOG Performance Status of 2 or less
7. Patient must not be on anti-retrovirals since they may alter patient metabolism

Exclusion Criteria:

1. Patient is not a candidate for definitive cancer surgery
2. Definitive cancer surgery can not be performed within 4-12 weeks post study enrollment as determined by the enrolling physician.
3. Body Mass Index < 21
4. Another malignancy within the past 6 months that was not a non-melanomatous skin lesion
5. ECOG Performance Status >2
6. Patient on anti-retrovirals since they may alter patient metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Change in miR-21 expression assessed in serum | Baseline up to 12 weeks
  Will be evaluated by a two-sided paired t-test at significance level 0.05.

SECONDARY OUTCOMES:
Overall adherence with diet intervention defined as 90% of all logged events meeting the diet restriction target | Up to 12 weeks
Change in body composition, assessed via BodyMetrix | Baseline up to 12 weeks
  Will be analyzed via a paired t-test.
Change in prostate tumor gene expression | Baseline up to 12 weeks
Change in weight, defined as a percent change | Baseline up to 12 weeks
  Will be assessed by modeling BMI as a function of time via mixed-effects regression.
Change in temperature | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in genomic expression of microRNA 21 (miR-21) | Baseline to after definitive surgery
  Initial cancer biopsy specimen for genomic analysis will be comped to definitive surgical specimens.
Change in insulin | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in biome analysis assessed by rectal swab | Baseline to 12 weeks
Change in psycho-social outcomes, assessed by the FACT-B | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Changes in nutritional status assessed by a Mini Nutritional Assessment (MNA) | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Local recurrence, assessed through patient records | From the date of study enrollment to time of event, assessed up to 12 weeks
  Will be analyzed via survival methods, specifically the Kaplan-Meier method and the log-rank test. If sufficient events occur, may assess the impact of various patient and clinical/treatment variables on these outcomes via Cox proportional hazards regression. Will be assessed and compared with historic controls using the Kaplan Meier method.
Distant metastases, assessed through patient records | From the date of study enrollment to time of event, assessed up to 12 weeks
  Will be analyzed via survival methods, specifically the Kaplan-Meier method and the log-rank test. If sufficient events occur, may assess the impact of various patient and clinical/treatment variables on these outcomes via Cox proportional hazards regression. Will be assessed and compared with historic controls using the Kaplan Meier method.
Progression free survival, assessed through patient records | From the date of study enrollment to time of event, assessed up to 12 weeks
  Will be analyzed via survival methods, specifically the Kaplan-Meier method and the log-rank test. If sufficient events occur, may assess the impact of various patient and clinical/treatment variables on these outcomes via Cox proportional hazards regression. Will be assessed and compared with historic controls using the Kaplan Meier method.
Overall survival, assessed through patient records | From the date of study enrollment to time of event, assessed up to 12 weeks
  Will be analyzed via survival methods, specifically the Kaplan-Meier method and the log-rank test. If sufficient events occur, may assess the impact of various patient and clinical/treatment variables on these outcomes via Cox proportional hazards regression. Will be assessed and compared with historic controls using the Kaplan Meier method.
Change in weight, defined by body mass index as weight in kg divided by height in meters squared | Baseline up to 12 weeks
  Will be assessed by modeling BMI as a function of time via mixed-effects regression.
Change in blood pressure | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in heart rate | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in respiratory rate | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in psycho-social outcomes, assessed by the FACT-P | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in psycho-social outcomes, assessed by the FACT-En | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.
Change in psycho-social outcomes, assessed by the POMIS cancer fatigue short form | Baseline up to 12 weeks
  Will be assessed as a function of time via mixed-effects regression.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/